CLINICAL TRIAL: NCT06460103
Title: Effect of Implant Surface Hydrophilicity on Peri-Implant Bone Formation Around Simultaneously Grafted Transiently Placed Titanium Zirconium Dental Small Diameter Implants - A Randomized Controlled Human Histometric Clinical Trial
Brief Title: Peri-implant Bone Formation of Grafted Sites Around Hydrophilic and Non-hydrophilic Dental Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Alexandre Perez, Head of Oral surgery and implantology unit, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AP2022-06
Record Dates: First submitted 2024-05-28; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Partially Edentulous Maxilla; Partially Edentulous Mandible
Keywords: Dental implants; SLActive; Hydrophile surface

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treatment blinding will not be possible as both device types, i.e. test and control implants, can be easily visually differentiated during handling and implantation. Test and control groups will be blinded for evaluation and statistical analysis and performed by independent laboratories.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Straumann® Bone Level Tapered SLActive®" mini-implant (hydrophilic surface) (Experimental): Tooth extraction + "Straumann® Bone Level Tapered, SLActive®" mini-implant placement + bone augmentation (bone graft "maxgraft® cortico-cancellous granules 0.5-2.0mm" and dental membrane "collprotect®membrane")
  Interventions: Device: Placement of a "Straumann® Bone Level Tapered implant SLActive®" (hydrophilic surface)
- "Straumann® Bone Level Tapered implants SLA®" mini-implant (hydrophobic surface) (Active Comparator): Tooth extraction + "Straumann® Bone Level Tapered , SLA®" mini-implant placement + bone augmentation (bone graft "maxgraft® cortico-cancellous granules 0.5-2.0mm" and dental membrane "collprotect®membrane")
  Interventions: Device: Placement of a "Straumann® Bone Level Tapered implant SLA®" (hydrophobic surface)

INTERVENTIONS:
Device: Placement of a "Straumann® Bone Level Tapered implant SLActive®" (hydrophilic surface) — Immediately after tooth extraction, patients will receive a "Straumann® Bone Level Tapered SLActive®" mini-implant at the ideal prosthetic position of the final implant, and bone augmentation using bone graft "maxgraft® " and dental membrane "collprotect®membrane".
  The mini-implant will be removed as a core trephine biopsy; the resulting osteotomies will be fine-prepared, and the final permanent implant will be placed after a healing period of 3 weeks post-augmentation.
  Arms: "Straumann® Bone Level Tapered SLActive®" mini-implant (hydrophilic surface)
Device: Placement of a "Straumann® Bone Level Tapered implant SLA®" (hydrophobic surface) — Immediately after tooth extraction, patients will receive a "Straumann® Bone Level Tapered SLA®" mini-implant at the ideal prosthetic position of the final implant, and bone augmentation using bone graft "maxgraft® " and dental membrane "collprotect®membrane".
  The mini-implant will be removed as a core trephine biopsy; the resulting osteotomies will be fine-prepared, and the final permanent implant will be placed after a healing period of 3 weeks post-augmentation.
  Arms: "Straumann® Bone Level Tapered implants SLA®" mini-implant (hydrophobic surface)

SUMMARY:
Although bone grafting at the same time as the placement of dental implants is a common procedure in implantology, there are currently no data on the influence of different types of implant surfaces on bone healing, which is crucial for implant stability.

The primary objective of this study is to assess if implant surface properties, i.e. hydrophilicity, affect the osseointegration of the implant in simultaneously augmented bone.

The secondary objective is to assess if implant surface properties, i.e. surface hydrophilicity, may affect the quantity of newly formed bone in the implant in simultaneously augmented bone.

Surface hydrophilicity modification is a well-adapted concept in dental implantology and is clinically well-established.

In this prospective study, all participants will receive a bone graft after extraction. After randomization, one group will receive a provisional SLA surface implant and another group will receive a provisional SLActive surface implant. The same standard surgical procedure will be performed for both groups when the definitive implant will be placed.

The study will run for a total of 3 year, and 35 patients per group will be included.

The Straumann SLA and SLActive implants, Maxgraft allograft and collprotect collagen membranes used in this study are all approved products on the Swiss market.

DETAILED DESCRIPTION:
The proposed study aims to histometrically investigate the influence of Titanium dental implant surface properties on the peri-implant bone formation in simultaneously bone-augmented implantation sites.

The magnitude of peri-implant bone formation and implant integration in augmented bone are clinically relevant for various clinical success criteria, including, e.g. long-term mechanical and aesthetic stability of load-bearing dental implants. Implant integration in simultaneously augmented bone, i.e. the investigated indication, can be considered critical for the success of approx. 40 to 50 % of all performed dental implant procedures world wide. The investigated subject is believed to be directly clinically relevant.

A common strategy to promote implant osseointegration and long-term implant stability is based on modifying Titanium dental implant surfaces' topographical and physicochemical properties.

The influence of topographical and physicochemical surface properties, including surface energy and hydrophilicity, of dental implants on the rate and extend of osseointegration in native bone has been well described. Also, the physicochemical material characteristics of bone substitutes have been shown to influence the rate of bone formation in augmented sites. Despite this thorough understanding of the individual influences of implant and bone graft properties, the interaction and synergistic properties between Titanium and Titanium Zirconium dental implant surfaces and bone substitutes on dental implant integration and bone formation in augmented sites remain widely undocumented. Investigations on a possible influence of implant surface/bone graft combination on implant osseointegration and peri-implant bone formation remain limited to very defined animal model systems. It is currently unclear if the preclinically observed effects may translate and be valid for human subjects. Consequently, the proposed study hypotheses that implant surface hydrophilicity may influence implant osseointegration and peri-implant bone formation in simultaneously augmented sites is novel, clinically undocumented, whilst highly relevant for the clinical and aesthetic success of a relevant portion of dental implant procedures.

The investigation is planned to be performed in patients displaying single hopeless teeth diagnosed for extraction and replacement by single implants requiring prior bone augmentation at the extraction site. The placement and retrieval of mini-implants are not considered to increase the number or significantly impact the type of planned interventions compared to routine treatment.

Specifically, treatments for the described indication consist of a 2-staged procedure requiring extraction and bone augmentation (first stage) followed by a second procedure for implant placement (second stage). The proposed study's design will be based on the placement of a mini implant in the centre of the extraction site as part of the first augmentation procedure. The mini-implant placement does not affect the treatment plan or outcome. It does not expose the patients to additional risks compared to routine treatment. By contrast, mini-implant placement may help reduce any potential risks for graft displacement of the bone augmentation and may support bone formation within the augmented area.

The second stage procedure will be used to retrieve the mini-implant using a core biopsy trephine instead of preparing the osteotomy by conventional drilling. The resulting osteotomy will be subsequently fine-prepared for the final, permanent implant placement. The required exact placement of the mini-implant at the planned ideal prosthetic position of the final implant can be considered routine, is clinically well-plannable and can be well-controlled as part of the available modern treatment workflows. The treatment sequence and outcome for the patient, i.e. a permanent implant-born restoration, is not expected to be affected by the planned investigation-related intervention, i.e. the placement and retrieval of a mini-implant.

From a parametric and methodological standpoint, histometric analysis can be considered the method of choice to study and quantify bone-to-implant contact and peri-implant bone formation. The patients will be recruited from regular patients diagnosed according to the described indication and scheduled for treatment at the University Hospital of Geneva.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Patients with a diagnosed indication for single tooth extraction and scheduled for consented replacement by an implant-based restoration requiring prior bone augmentation
* Only patients displaying periodontally healthy teeth adjacent to the extracted teeth shall be included (probing depth (PD) < 4mm, no bleeding on probing (BOP)
* Patients must be physically and psychologically able to undergo implant surgery and restorative procedures (American Academy of Anesthesiologist class I or II)

Exclusion Criteria:

* Presence of any general contra-indication related to implant therapy
* Heavy smokers ( ≥10 cigarettes/day)
* Patients displaying a history of uncontrolled metabolic disorders (e.g. diabetes mellitus)
* Patients with a history of malignancy, radiotherapy, or chemotherapy
* Pregnant or breast feeding patients
* Patients with a history of immunodeficiencies
* Patients displaying any metabolic bone disease
* Patients with disturbed bone or wound healing
* Patients with untreated or active periodontitis (BOP and PD>5mm)
* Extraction sites displaying an absent or defections buccal bone plate
* Vulnerable patients will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Bone-to-Implant Contact (BIC) | 3 weeks after implant placement
  The cross-sectional implant perimeter percentage in direct contact with newly formed bone over the total cross-sectional implant perimeter. Only the perimeter in contact with augmented bone will be considered for measuring this parameter.

SECONDARY OUTCOMES:
Percentage of newly formed bone area | 3 weeks after implant placement
  The histological cross-sectional area covered by newly formed bone over the total cross-sectional area within a defined region of interest within the augmented sites.
Graft particle area | 3 weeks after implant placement
  The histological cross-sectional area covered by remaining graft particles over the total cross-sectional area within a defined region of interest within the augmented sites.
Assessment of the tissue inflammatory response | 3 weeks after implant placement
  A region of interest within the histological cross-sections of augmented areas will be evaluated with regards to the inflammatory tissue response by quantifying the number of white blood cells to determine the inflammatory score using a standardized four-point scoring scale ranging from "-" for not present to "+++" for markedly present.
Assessment of the healing response | 3 weeks after implant placement
  Vascularization, osteoblasts, and osteoclasts will be scored using a standardized four-point scoring scale ranging from "-" for not present to "+++" for markedly present.This measure will be used to assess the implant surface/bone graft combination's overall healing reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Perez, Dr, Principal Investigator — University of Geneva